CLINICAL TRIAL: NCT03484923
Title: A Randomized, Open-label, Phase II Open Platform Study Evaluating the Efficacy and Safety of Novel Spartalizumab (PDR001) Combinations in Previously Treated Unresectable or Metastatic Melanoma
Brief Title: Study of Efficacy and Safety of Novel Spartalizumab Combinations in Patients With Previously Treated Unresectable or Metastatic Melanoma
Acronym: PLATforM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001J2201; 2018-000610-38 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
Keywords: Unresectable; melanoma; metastatic melanoma; advanced melanoma; spartalizumab; PDR001; LAG525; capmatinib; INC280; canakinumab; ACZ885; ribociclib; LEE011; immunotherapy; platform study; LAG-3
MeSH Terms: conditions — Melanoma | interventions — spartalizumab; capmatinib; canakinumab; ribociclib

STUDY DESIGN:
Masking Description: After approval of protocol amendment 5 (26Jun2020), a non-randomized single arm was added
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: LAG525 + PDR001 (randomized section) (Experimental): Participnats randomized to receive LAG525 at a dosage of 600 mg administered intravenously every 4 weeks, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
  Interventions: Drug: PDR001; Drug: LAG525
- Arm 2: INC280+PDR001 (randomized section) (Experimental): Participants randomized to receive INC280 orally at a dosage of 400 mg twice daily, in combination with PDR001 intravenously at a dosage of 400 mg every 4 weeks
  Interventions: Drug: PDR001; Drug: INC280
- Arm 3: ACZ885 + PDR001 (randomized section) (Experimental): Participants randomized to receive to receive ACZ885 at a dosage of 300 mg administered subcutaneously every 4 weeks, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
  Interventions: Drug: PDR001; Drug: ACZ885
- Arm 4: LEE011 + PDR001 (randomized section) (Experimental): Participants randomized to receive LEE011 orally at a dosage of 600 mg once daily on Days 1-21 of a 28-day cycle, in combination with PDR001 intravenously at a dosage of 400 mg every 4 weeks
  Interventions: Drug: PDR001; Drug: LEE011
- Arm 1A: LAG525 + PDR001 (non-randomized section) (Experimental): LAG-3 positive participants received LAG525 at a dosage of 600 mg administered intravenously every 4 weeks, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
  Interventions: Drug: PDR001; Drug: LAG525

INTERVENTIONS:
Drug: PDR001 — 400 mg of PDR001 administered every 4 weeks intravenously
  Other Names: Spartalizumab
Drug: LAG525 — 600 mg of LAG525 administered every 4 weeks intravenously
  Other Names: Ieramilimab
  Arms: Arm 1: LAG525 + PDR001 (randomized section); Arm 1A: LAG525 + PDR001 (non-randomized section)
Drug: INC280 — 400 mg of INC280 administered twice daily orally
  Other Names: Capmatinib
  Arms: Arm 2: INC280+PDR001 (randomized section)
Drug: ACZ885 — 200 mg of ACZ885 administered every 4 weeks subcutaneosuly
  Other Names: Canakinumab
  Arms: Arm 3: ACZ885 + PDR001 (randomized section)
Drug: LEE011 — 600 mg of LEE011 orally taken once daily on Days 1-21 of a 28-day cycle
  Other Names: Ribociclib
  Arms: Arm 4: LEE011 + PDR001 (randomized section)

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of novel spartalizumab (PDR001) combinations in previously treated unresectable or metastatic melanoma

DETAILED DESCRIPTION:
This study was a randomized, open-label, two-part, multi-center, open platform phase II study designed to evaluate the efficacy and safety of the anti-PD-1 antibody PDR001 in combination with novel agents for previously treated unresectable or metastatic melanoma. Additionally, a non-randomized single-arm was added based on interim analysis findings to assess the efficacy and safety of PDR001 in combination with LAG525 in subjects with previously treated unresectable or metastatic LAG-3 positive melanoma.

The study consisted of two parts: the selection part and the expansion part, which were applicable to both the randomized and non-randomized sections. In the randomized section, participants were randomized to one of four combination arms available for enrollment:

* Arm 1: LAG525 600 mg intravenously (i.v.) every 4 weeks (Q4W) and PDR001 400 mg i.v. Q4W.
* Arm 2: INC280 400 mg orally (p.o.) twice daily (BID) and PDR001 400 mg i.v. Q4W.
* Arm 3: ACZ885 300 mg subcutaneously (s.c.) every 4 weeks (Q4W) and PDR001 400 mg i.v. Q4W.
* Arm 4: LEE011 600 mg p.o. once daily (QD) on Days 1-21 of a 28-day cycle and PDR001 400 mg i.v. Q4W.

At each interim analysis, the following determinations were made: (1) which arm met the pre-specified efficacy criteria and expanded to the expansion part, (2) which arms continued enrollment in selection part (up to 45 subjects), and (3) which arms were discontinued due to futility, considering efficacy, safety, and biomarker data. The expansion phase included enrollment of subjects only in the combination arms that met the pre-specified criteria in selection part.

In the non-randomized section, a single combination arm was opened for enrollment in selection part:

• Arm 1A: LAG525 600 mg i.v. Q4W and PDR001 400 mg i.v. Q4W, assessed in a population selected based on the LAG-3 status of their tumor.

Arm 1A would be eligible for enrollment in expansion part only if it met the pre-specified criterion for this arm.

Participants received the study treatment corresponding to their assigned arm on a 28-day cycle basis until disease progression, as determined by local assessment using RECIST v1.1 criteria, or until certain events occurred, such as unacceptable toxicity, initiation of subsequent anti-cancer therapy, withdrawal of consent, investigator's decision, loss to follow-up, death, or termination of the study by the sponsor. Following discontinuation of the study treatment, all subjects were monitored for safety evaluations for up to 150 days after their last dose of the study treatment.

ELIGIBILITY:
Key inclusion criteria for Arm 1, 2, 3, 4:

* Histologically confirmed unresectable or metastatic stage IIIB/C/D or IV melanoma using AJCC edition 8.
* Previously treated for unresectable or metastatic melanoma:

  * Subjects with V600BRAF wild-type disease had to have received prior systemic therapy for unresectable or metastatic melanoma with anti-PD-1/PD-L1. Additionally, subjects may have received anti-CTLA-4 as a single agent or in combination with anti-PD-1/PD-L1, irrespective of the sequence. No additional systemic treatment was allowed for advanced or metastatic melanoma.

A maximum of two prior lines of systemic therapies for unresectable or metastatic melanoma were allowed.

The last dose of prior therapy (anti-PD-1, anti-PD-L1, or anti-CTLA-4) had to have been received more than four weeks before randomization.

* Subjects with V600BRAF mutant disease had to have received prior systemic therapy for unresectable or metastatic melanoma with anti-PD-1/PD-L1 and V600BRAF inhibitor. Additionally, subjects may have received anti-CTLA-4 as a single agent or in combination with anti-PD-1/PD-L1, or MEK inhibitor (in combination with V600BRAF inhibitor or as a single agent), irrespective of the sequence. No additional systemic treatment was allowed for advanced or metastatic melanoma.
* A maximum of three prior lines of systemic therapies for unresectable or metastatic melanoma were allowed.
* The last dose of prior therapy had to have been received more than 4 weeks (for anti-PD-1, anti-PD-L1, or anti-CTLA-4) or more than 2 weeks (for V600BRAF or MEK inhibitor) prior to randomization.
* All subjects (with V600BRAF wild-type disease and with V600BRAF mutant disease) had to have documented disease progression as per RECIST v1.1 while on/after the last therapy received prior to study entry and while on/after treatment with anti-PD1/PD-L1. The last progression had to have occurred within 12 weeks prior to randomization in the study.

  * ECOG performance status 0-2.
  * At least one measurable lesion per RECIST v1.1.
  * At least one lesion, suitable for sequential mandatory tumor biopsies (screening and on-treatment) in accordance with the biopsy guidelines specified in the protocol. The same lesion had to be biopsied sequentially.
  * Screening tumor biopsy had to fulfill the tissue quality criteria outlined in the protocol, as assessed by a local pathologist.

Key inclusion criteria for Arm 1A:

* Histologically confirmed unresectable or metastatic stage IIIB/C/D or IV melanoma according to AJCC Edition 8.
* Previously treated for unresectable or metastatic melanoma:

  * All subjects had to have received anti-PD-1 checkpoint inhibitor therapy (i.e., pembrolizumab or nivolumab) either as monotherapy or in combination with ipilimumab as the last systemic therapy prior to enrollment and had to have confirmed disease progression as per RECIST v1.1 (confirmed on a subsequent scan, which could be the scan performed during screening) while on or after this therapy prior to enrollment.
  * Subjects with V600BRAF wild-type disease had to have received no more than 2 prior systemic therapies, including prior anti-PD-1/PD-L1 (as monotherapy or in combination with ipilimumab).
  * Subjects with V600BRAF mutant disease had to have received no more than 3 prior systemic therapies, including anti-PD-1/PD-L1 (as monotherapy or in combination with ipilimumab) and V600BRAF inhibitor (as monotherapy or in combination with a MEK inhibitor).
  * The last dose of anti-PD-1-based therapy had to have been received more than four weeks prior to the first dose of study treatment.
  * The last documented disease progression had to have occurred within 12 weeks prior to the first dose of study treatment.
  * No additional systemic treatment was allowed for advanced or metastatic melanoma (this included, for example, tumor-infiltrating lymphocyte therapy).
* ECOG performance status 0-1.
* At least one measurable lesion per RECIST v1.1.
* Subjects had to have a baseline tumor sample that was positive for LAG-3 per central assessment.

Key exclusion criteria common to all combination arms:

* Subjects with uveal or mucosal melanoma.
* Presence of clinically active or unstable brain metastasis at the time of screening.
* Use of any live vaccines against infectious diseases within 3 months before randomization/enrollment.
* Active infection requiring systemic antibiotic therapy at the time of randomization/enrollment.
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization/enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, were permitted in the absence of active autoimmune disease.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease.
* Prior allogenic bone marrow or solid organ transplant.
* History of known hypersensitivity to any of the investigational drugs used in this study.
* Malignant disease, other than that being treated in this study.
* Prior systemic therapy for unresectable or metastatic melanoma with any investigational agent or with any other agent except anti-PD-1/PD-L1 and anti-CTLA-4 (and V600BRAF and MEK inhibitors if the subject has V600BRAF mutant disease). Prior neoadjuvant and/or adjuvant therapy for melanoma completed less than 6 months before the start of the study treatment.
* Medical history or current diagnosis of myocarditis.
* Cardiac Troponin T (or Troponin I) level > 2 x ULN at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (6):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - UCSF Medical Center ., San Francisco, California
  - Massachusetts General Hospital Massachusetts Gen. Hospital CC, Boston, Massachusetts
  - NYU Laura and Isaac Perlmutter Cancer Center Perlmutter Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, München
- Italy (3):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: None of the arms were opened in the extension part.
Pre-assignment Details: The screening period began once written informed consent was provided and ended after 28 days (or after 35 days for subjects screened for Arm 1A) or when subject was randomized/enrolled, whichever came first. 1 participant randomized to Arm 3 discontinued before study treatment due to an AE.
Groups:
- Arm 1: LAG525 + PDR001 (Randomized Section): Participants randomized to receive LAG525 at a dosage of 600 mg administered intravenously every 4 weeks, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
- Arm 2: INC280+PDR001 (Randomized Section): Participants randomized to receive INC280 orally at a dosage of 400 mg twice daily, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
- Arm 3: ACZ885 + PDR001 (Randomized Section): Participants randomized to receive ACZ885 at a dosage of 300 mg administered subcutaneously every 4 weeks, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
- Arm 4: LEE011 + PDR001 (Randomized Section): Participants randomized to receive LEE011 orally at a dosage of 600 mg once daily on Days 1-21 of a 28-day cycle, in combination with PDR001 at a dosage of 400 mg administered intravenously every 4 weeks
Period: Overall Study
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Started | 45 | 43 | 43 | 44 | 21
Treated | 45 | 43 | 42 | 44 | 21
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 45 | 43 | 43 | 44 | 21
Not completed — Adverse Event | 3 | 3 | 5 | 11 | 1
Not completed — Death | 2 | 2 | 3 | 0 | 1
Not completed — Physician Decision | 6 | 7 | 6 | 3 | 2
Not completed — Progressive disease | 33 | 28 | 26 | 30 | 16
Not completed — Subject Decision | 1 | 3 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section) | Total
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 28 | 28 | 8 | 122
  >=65 years | 16 | 14 | 15 | 16 | 13 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 15 | 14 | 9 | 76
  Male | 28 | 22 | 28 | 30 | 12 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 45 | 42 | 38 | 42 | 20 | 187
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 4 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the percentage of patients with a best overall response of either confirmed complete response (CR) or partial response (PR) as per local review by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and assessed by computed tomography (CT)/ magnetic resonance imaging (MRI).
  CR:Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 49 months (randomized section) and 18 months (non-randomized section)
Population: Randomized section: All participants to whom study treatment was assigned by randomization.
  Non-randomized section: All participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21
Percentage of participants | 8.9 [2.5 to 21.2] | 4.7 [0.6 to 15.8] | 4.7 [0.6 to 15.8] | 6.8 [1.4 to 18.7] | 14.3 [3.0 to 36.3]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the time from date of first documented CR or PR to date of first documented disease progression (as per local review by RECIST v1.1 and assessed by CT/MRI) or death due to any cause. Subjects continuing without progression or death due to underlying cancer were censored at the date of their last adequate tumor assessment.
  CR:Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first documented response to disease progression or death due to any cause, whichever occurs first, assessed up to 49 months (randomized part) and 18 months (non-randomized part)
Population: Randomized section: All participants to whom study treatment was assigned by randomization for whom best overall response was complete response or partial response.
  Non-randomized section: All participants who received at least one dose of study treatment for whom best overall response was complete response or partial response
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 4 | 2 | 2 | 3 | 3
Days | 476 [169 to 1373] | 941.5 [504 to 1379] | 617.5 [113 to 1122] | 217 [169 to 281] | 281 [169 to 449]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization (or date of first dose of study treatment in non-randomized part) to date of death due to any cause. The OS distribution was estimated using the Kaplan-Meier method, and the medians and 95% confidence intervals of the medians were presented.
Time Frame: From randomization (or start of treatment for non-randomized section) to death due to any cause, assessed up to 49 months (randomized section) and 24 months (non-randomized section)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21
Months | 8.8 [6.3 to 21.4] | 12.1 [6.6 to 18.5] | 8.7 [5.7 to 17.9] | 10.1 [7.4 to 15.6] | 14.0 [8.4 to NA] — NA: Not estimable due to the insufficient number of participants with events

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time between the date of randomization (or date of first dose of study treatment in non-randomized section) to the date of event defined as the first documented disease progression (as per local review by RECIST v1.1 and assessed by CT/MRI) or death due to any cause. If a subject had not had an event before leaving study or initiation of subsequent anticancer therapy, PFS was censored at the date of last adequate tumor assessment. The PFS distribution was estimated using the Kaplan-Meier method, medians and 95% confidence interval of the medians were presented.
Time Frame: From randomization (or start of treatment for non-randomized section) to disease progression or death due to any cause, whichever occurs first, assessed up to 49 months (randomized section) and 18 months (non-randomized section)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21
Months | 2.7 [1.7 to 2.8] | 2.7 [2.4 to 2.8] | 2.7 [2.6 to 2.8] | 2.8 [2.7 to 4.4] | 2.8 [2.7 to 4.6]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with best overall response of CR, PR or stable disease (SD) (as per local review by RECIST v1.1 and assessed by CT/MRI).
  CR:Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to 49 months (randomized section) and 18 months (non-randomized section)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21
Percentage of participants | 15.6 [6.5 to 29.5] | 16.3 [6.8 to 30.7] | 18.6 [8.4 to 33.4] | 31.8 [18.6 to 47.6] | 33.3 [14.6 to 57.0]

6. Secondary Outcome: Percentage of Participants With PDR001 Anti-drug Antibodies (ADA) Positive Result at Baseline
Description: Percentage of participants who had a PDR001 ADA positive result at baseline.
Time Frame: At Baseline
Population: Randomized section: Participants to whom study treatment was assigned by randomization with a determinant baseline immunogenicity sample for PDR001.
  Non-randomized section: Participants who received at least one dose of treatment with a determinant baseline immunogenicity sample for PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 43 | 38 | 40 | 41 | 20
Participants | 1 | 0 | 1 | 0 | 0

7. Secondary Outcome: Percentage of Participants With LAG525 Anti-drug Antibodies (ADA) Positive Result at Baseline
Description: Percentage of participants who had a LAG525 ADA positive result at baseline. Only applicable for participants enrolled in Arm 1 and Arm 1A.
Time Frame: At Baseline
Population: Randomized section: Participants randomized to Arm 1 with a determinant baseline immunogenicity sample for LAG525.
  Non-randomized section: Participants who received at least one dose of treatment with a determinant baseline immunogenicity sample for LAG525.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 43 | 20
Participants | 3 | 0

8. Secondary Outcome: Percentage of Participants With ACZ885 Anti-drug Antibodies (ADA) Positive Result at Baseline
Description: Percentage of participants who had an ACZ885 ADA positive result at baseline. Only applicable for subjects enrolled in Arm 3.
Time Frame: At Baseline
Population: Participants randomized to Arm 3 with a determinant baseline immunogenicity sample for ACZ885.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: ACZ885 + PDR001 (Randomized Section)
Number analyzed (Participants) | 39
Participants | 0

9. Secondary Outcome: Percentage of Participants Who Were Treatment-induced ADA Positive and Treatment-boosted ADA Positive for PDR001
Description: Percentage of participants who tested positive for treatment-induced ADA for PDR001 (subjects with ADA-negative sample at baseline with at least one post-baseline ADA positive sample) as well as treatment-boosted ADA for PDR001 (subjects with baseline positive ADA titre that was boosted to a 4-fold or higher-level following treatment).
Time Frame: Pre-infusion on Day 1 of Cycle 1, 2, 3, 4, 5, 6 and thereafter every 3 cycles until end of treatment (EOT), EOT, and 30 and 150 days post-EOT (assessed up to 49 months randomized section and 24 months non-randomized section). Cycle= 28 days
Population: Randomized section: Participants to whom study treatment was assigned by randomization with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample.
  Non-randomized section: Participants who received at least one dose of study treatment with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 40 | 34 | 38 | 39 | 19
Participants | 3 | 5 | 3 | 0 | 0

10. Secondary Outcome: Percentage of Participants Who Were Treatment-induced ADA Positive and Treatment-boosted ADA Positive for LAG525
Description: Percentage of participants who tested positive for treatment-induced ADA for LAG525 (subjects with ADA-negative sample at baseline with at least one post-baseline ADA positive sample) as well as treatment-boosted ADA for LAG525 (subjects with baseline positive ADA titre that was boosted to a 4-fold or higher-level following treatment). Only applicable for subjects enrolled in Arm 1 and Arm 1A.
Time Frame: Pre-infusion on Day 1 of Cycle 1, 2, 3, 4, 5, 6 and thereafter every 3 cycles until end of treatment (EOT) and EOT (assessed up to 49 months in the randomized section and 18 months in the non-randomized section). Cycle= 28 days
Population: Randomized section: Participants randomized to Arm 1 with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample.
  Non-randomized section: Participants who received at least one dose of study treatment with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 40 | 19
Participants | 7 | 2

11. Secondary Outcome: Percentage of Participants Who Were Treatment-induced ADA Positive and Treatment-boosted ADA Positive for ACZ885
Description: Percentage of participants who tested positive for treatment-induced ADA for ACZ885 (subjects with ADA-negative sample at baseline with at least one post-baseline ADA positive sample) as well as treatment-boosted ADA for ACZ885 (subjects with baseline positive ADA titre that was boosted to a 4-fold or higher-level following treatment). Only applicable for subjects enrolled in Arm 3.
Time Frame: Pre-infusion on Day 1 of Cycle 1, 2, 3, 4, 5, 6 and thereafter every 3 cycles until end of treatment (EOT) and EOT (assessed up to 40 months). Cycle= 28 days
Population: Participants randomized to Arm 3 with a determinant baseline immunogenicity sample and at least one determinant post-baseline immunogenicity sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: ACZ885 + PDR001 (Randomized Section)
Number analyzed (Participants) | 38
Participants | 1

12. Secondary Outcome: Percentage of Participants With a Favorable Biomarker Profile (pFBP)
Description: Biomarker parameters included: 1) number of tumor infiltrating T cells (TIL), 2) activation level of TIL, and 3) changes in immune response gene expression signatures. For the number of TILs, an increase in tumoral CD8+ cell numbers compared to baseline was considered favorable. The activation level of TIL was assessed by the percentage of tumoral CD8+ cells expressing GzmB (a marker for cytotoxic activity) or Ki67 (a marker for cell proliferation), where an increase in either GZMB+/CD8+ or KI67+/CD8+ post-baseline was considered favorable. Changes in immune response gene expression signatures were evaluated by the levels in T-cell inflamed signature (TIS), where an increase from baseline was considered favorable.
  To be categorized as having a pFBP, a subject must meet the favorable criteria for at least two of the three biomarker parameters. The percentage of participants with pFBP was assessed.
Time Frame: Baseline and after 3-4 weeks of treatment
Population: Participants who received at least one dose of treatment with an evaluable baseline tumor biopsy sample and at least one evaluable post-baseline tumor biopsy sample with evaluable results for the three biomarker parameters.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 22 | 21 | 31 | 6 | 0
Percentage of participants | 13.6 [2.9 to 34.9] | 4.8 [0.1 to 23.8] | 6.5 [0.8 to 21.4] | 16.7 [0.4 to 64.1] |

13. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment: deaths collected from day of patient's informed consent to the day before the first administration of study treatment.
  On-treatment: deaths collected from start of treatment to 30 days after last dose of study treatment.
  Extended safety follow-up: deaths collected from 31 days after last dose of study treatment up to 150 days after last dose of PDR001 (if this timepoint was later than 30 days after last dose of study treatment) Post-treatment survival follow-up: deaths collected from day 151 post-last dose of PDR001 or 31 days after last dose of study treatment (whichever occurred last) up to end of study.
Time Frame: Pre-treatment: up to 28/35 days (randomized/non-randomized). On-treatment: up to 49/19 months (randomized/non-randomized). Extended safety FU and Post-treatment survival FU: up to 49/24 months (randomized/non-randomized).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Section) | Arm 2: INC280+PDR001 (Randomized Section) | Arm 3: ACZ885 + PDR001 (Randomized Section) | Arm 4: LEE011 + PDR001 (Randomized Section) | Arm 1A: LAG525 + PDR001 (Non-randomized Section)
Number analyzed (Participants) | 45 | 43 | 43 | 44 | 21
Participants
  Pre-treatment deaths | 0 | 0 | 0 | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 45 | 43 | 42 | 44 | 21
  On-treatment deaths | 5 | 3 | 3 | 3 | 1
  Extended safety follow-up deaths: number analyzed (Participants) | 45 | 43 | 42 | 44 | 21
  Extended safety follow-up deaths | 14 | 11 | 15 | 11 | 4
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 26 | 29 | 24 | 30 | 14
  Post-treatment survival follow-up deaths | 18 | 19 | 15 | 19 | 7
  All deaths | 37 | 33 | 33 | 33 | 12

ADVERSE EVENTS:
Time Frame: On-treatment: from first dose to 30 days post-treatment, up to 49/24 months (randomized/non-randomized) Extended safety follow-up: from 31 days after last dose of treatment up to 150 days after last dose of PDR001 (if >30 days post-treatment), up to 49/24 months (randomized/non-randomized) Post-treatment survival follow-up: from day 151 after last dose of PDR001 or 31 days post-treatment (whichever occurred last) up to end of study, up to 49/24 months (randomized/non-randomized).
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered AEs. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period. Safety analyses were performed in the safety set, including all participants who received at least one dose of treatment
Groups:
- Arm 1: LAG525 + PDR001 (Randomized Part)- On-treatment Period; Arm 2: INC280+PDR001 (Randomized Part)- On-treatment Period; Arm 3: ACZ885 + PDR001 (Randomized Part)- On-treatment Period; Arm 4: LEE011 + PDR001 (Randomized Part)- On-treatment Period; Arm 1A: LAG525 + PDR001 (Non-randomized Part)- On-treatment Period: AEs collected during on-treatment period (up to 30 days post-treatment)
- Arm 1: LAG525 + PDR001 (Randomized Part)- Extended Safety Follow-up; Arm 2: INC280+PDR001 (Randomized Part) - Extended Safety Follow-up; Arm 3: ACZ885 + PDR001 (Randomized Part)- Extended Safety Follow-up; Arm 4: LEE011 + PDR001 (Randomized Part)- Extended Safety Follow-up; Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Extended Safety Follow-up: AEs collected during extended safety follow-up period (from day 31 post-treatment up to 150 days post last dose of PDR001 [if >30 days post-treatment])
- Arm 1: LAG525 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up; Arm 2: INC280+PDR001 (Randomized Part)- Post-treatment Survival Follow-up; Arm 3: ACZ885 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up; Arm 4: LEE011 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up; Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Post-treatment Survival Follow-up: Deaths collected in the post- treatment survival follow-up period (starting from day 151 post- treatment). No AEs were collected during this period
Arm/Group | Arm 1: LAG525 + PDR001 (Randomized Part)- On-treatment Period | Arm 1: LAG525 + PDR001 (Randomized Part)- Extended Safety Follow-up | Arm 1: LAG525 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up | Arm 2: INC280+PDR001 (Randomized Part)- On-treatment Period | Arm 2: INC280+PDR001 (Randomized Part) - Extended Safety Follow-up | Arm 2: INC280+PDR001 (Randomized Part)- Post-treatment Survival Follow-up | Arm 3: ACZ885 + PDR001 (Randomized Part)- On-treatment Period | Arm 3: ACZ885 + PDR001 (Randomized Part)- Extended Safety Follow-up | Arm 3: ACZ885 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up | Arm 4: LEE011 + PDR001 (Randomized Part)- On-treatment Period | Arm 4: LEE011 + PDR001 (Randomized Part)- Extended Safety Follow-up | Arm 4: LEE011 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- On-treatment Period | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Extended Safety Follow-up | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Post-treatment Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 5/45 | 14/45 | 18/26 | 3/43 | 11/43 | 19/29 | 3/42 | 15/42 | 15/24 | 3/44 | 11/44 | 19/30 | 1/21 | 4/21 | 7/14
Serious Adverse Events (participants affected / at risk) | 21/45 | 5/45 | 0/0 | 21/43 | 0/43 | 0/0 | 12/42 | 4/42 | 0/0 | 22/44 | 8/44 | 0/0 | 7/21 | 2/21 | 0/0
Other Adverse Events (participants affected / at risk) | 40/45 | 5/45 | 0/0 | 42/43 | 6/43 | 0/0 | 32/42 | 5/42 | 0/0 | 44/44 | 9/44 | 0/0 | 18/21 | 2/21 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: LAG525 + PDR001 (Randomized Part)- On-treatment Period (N=45) | Arm 1: LAG525 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=45) | Arm 1: LAG525 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 2: INC280+PDR001 (Randomized Part)- On-treatment Period (N=43) | Arm 2: INC280+PDR001 (Randomized Part) - Extended Safety Follow-up (N=43) | Arm 2: INC280+PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 3: ACZ885 + PDR001 (Randomized Part)- On-treatment Period (N=42) | Arm 3: ACZ885 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=42) | Arm 3: ACZ885 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 4: LEE011 + PDR001 (Randomized Part)- On-treatment Period (N=44) | Arm 4: LEE011 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=44) | Arm 4: LEE011 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- On-treatment Period (N=21) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Extended Safety Follow-up (N=21) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Myocarditis (Cardiac disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Adrenal haematoma (Endocrine disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 1 | NA | 1 | 0 | NA | 0 | 0 | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Gastritis (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Intussusception (Gastrointestinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Nausea (Gastrointestinal disorders) | 2 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Subileus (Gastrointestinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 1 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA
Asthenia (General disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Chest pain (General disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Fatigue (General disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 1 | NA | 0 | 0 | NA
General physical health deterioration (General disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA
Heteroplasia (General disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Oedema peripheral (General disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Pain (General disorders) | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Pyrexia (General disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 2 | NA | 0 | 0 | NA
Cholangitis (Hepatobiliary disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
Cytokine release syndrome (Immune system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Drug hypersensitivity (Immune system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Cellulitis (Infections and infestations) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Erysipelas (Infections and infestations) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Infection (Infections and infestations) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Pneumonia (Infections and infestations) | 0 | 2 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Pneumonia bacterial (Infections and infestations) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Respiratory tract infection (Infections and infestations) | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Sepsis (Infections and infestations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Skin infection (Infections and infestations) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Suspected COVID-19 (Infections and infestations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Ocular procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Blood lactic acid increased (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
General physical condition abnormal (Investigations) | 2 | 1 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA
Haemoglobin decreased (Investigations) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Liver function test abnormal (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Liver function test increased (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 2 | 1 | NA | 0 | 0 | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | NA | 1 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Dizziness (Nervous system disorders) | 0 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Epilepsy (Nervous system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Facial paresis (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Headache (Nervous system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hemiparesis (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Nervous system disorder (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Peripheral nerve paresis (Nervous system disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Seizure (Nervous system disorders) | 1 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Spinal cord compression (Nervous system disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA
Device dislocation (Product Issues) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Renal failure (Renal and urinary disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA | 0 | 0 | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 1 | NA | 0 | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Hypotension (Vascular disorders) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Peripheral ischaemia (Vascular disorders) | 0 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Phlebitis (Vascular disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Vena cava thrombosis (Vascular disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Venous thrombosis (Vascular disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: LAG525 + PDR001 (Randomized Part)- On-treatment Period (N=45) | Arm 1: LAG525 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=45) | Arm 1: LAG525 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 2: INC280+PDR001 (Randomized Part)- On-treatment Period (N=43) | Arm 2: INC280+PDR001 (Randomized Part) - Extended Safety Follow-up (N=43) | Arm 2: INC280+PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 3: ACZ885 + PDR001 (Randomized Part)- On-treatment Period (N=42) | Arm 3: ACZ885 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=42) | Arm 3: ACZ885 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 4: LEE011 + PDR001 (Randomized Part)- On-treatment Period (N=44) | Arm 4: LEE011 + PDR001 (Randomized Part)- Extended Safety Follow-up (N=44) | Arm 4: LEE011 + PDR001 (Randomized Part)- Post-treatment Survival Follow-up (N=0) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- On-treatment Period (N=21) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Extended Safety Follow-up (N=21) | Arm 1A: LAG525 + PDR001 (Non-randomized Part)- Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | NA | 6 | 1 | NA | 6 | 1 | NA | 11 | 0 | NA | 3 | 1 | NA
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | NA | 0 | 0 | NA | 1 | 1 | NA | 4 | 0 | NA | 0 | 0 | NA
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | NA | 2 | 0 | NA | 1 | 0 | NA | 7 | 0 | NA | 1 | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | NA | 0 | 0 | NA | 1 | 0 | NA | 20 | 0 | NA | 0 | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | NA | 1 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA
Hypothyroidism (Endocrine disorders) | 2 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 2 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | NA | 3 | 0 | NA | 5 | 0 | NA | 5 | 0 | NA | 2 | 0 | NA
Constipation (Gastrointestinal disorders) | 8 | 0 | NA | 6 | 1 | NA | 7 | 0 | NA | 3 | 1 | NA | 0 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | NA | 10 | 1 | NA | 3 | 0 | NA | 9 | 1 | NA | 5 | 0 | NA
Dry mouth (Gastrointestinal disorders) | 3 | 0 | NA | 1 | 0 | NA | 4 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA
Nausea (Gastrointestinal disorders) | 13 | 0 | NA | 18 | 0 | NA | 9 | 1 | NA | 15 | 2 | NA | 6 | 0 | NA
Vomiting (Gastrointestinal disorders) | 6 | 0 | NA | 11 | 0 | NA | 3 | 0 | NA | 8 | 1 | NA | 3 | 0 | NA
Asthenia (General disorders) | 9 | 1 | NA | 7 | 1 | NA | 7 | 0 | NA | 8 | 2 | NA | 7 | 0 | NA
Chest pain (General disorders) | 2 | 0 | NA | 3 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Chills (General disorders) | 1 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 1 | 0 | NA
Fatigue (General disorders) | 7 | 1 | NA | 5 | 0 | NA | 5 | 1 | NA | 8 | 1 | NA | 4 | 0 | NA
Oedema peripheral (General disorders) | 3 | 0 | NA | 10 | 0 | NA | 1 | 0 | NA | 3 | 0 | NA | 1 | 0 | NA
Pain (General disorders) | 4 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 2 | NA | 0 | 0 | NA
Pyrexia (General disorders) | 3 | 0 | NA | 13 | 0 | NA | 2 | 0 | NA | 8 | 2 | NA | 2 | 0 | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA
Rhinitis (Infections and infestations) | 3 | 0 | NA | 3 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | NA | 6 | 0 | NA | 2 | 1 | NA | 15 | 2 | NA | 1 | 0 | NA
Amylase increased (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 3 | 1 | NA | 1 | 0 | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | NA | 5 | 0 | NA | 3 | 0 | NA | 17 | 1 | NA | 1 | 0 | NA
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | NA | 2 | 0 | NA | 2 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
Blood creatinine increased (Investigations) | 0 | 0 | NA | 5 | 0 | NA | 1 | 0 | NA | 4 | 0 | NA | 0 | 0 | NA
Blood lactate dehydrogenase increased (Investigations) | 3 | 2 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
Blood potassium decreased (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | NA | 2 | 0 | NA | 1 | 0 | NA | 3 | 1 | NA | 0 | 0 | NA
Haemoglobin decreased (Investigations) | 1 | 0 | NA | 2 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 2 | 1 | NA
Lipase increased (Investigations) | 3 | 1 | NA | 3 | 0 | NA | 3 | 0 | NA | 5 | 0 | NA | 2 | 0 | NA
Neutrophil count decreased (Investigations) | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA
Platelet count decreased (Investigations) | 2 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
SARS-CoV-2 test negative (Investigations) | 0 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 4 | 1 | NA | 0 | 0 | NA
Weight decreased (Investigations) | 6 | 0 | NA | 2 | 0 | NA | 5 | 1 | NA | 4 | 2 | NA | 0 | 0 | NA
White blood cell count decreased (Investigations) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 4 | 0 | NA | 0 | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 10 | 0 | NA | 3 | 1 | NA | 7 | 0 | NA | 9 | 2 | NA | 2 | 0 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | 3 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | NA | 2 | 1 | NA | 2 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | NA | 4 | 0 | NA | 2 | 0 | NA | 6 | 0 | NA | 2 | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | NA | 3 | 2 | NA | 1 | 0 | NA | 3 | 1 | NA | 0 | 0 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 1 | 1 | NA | 2 | 0 | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | NA | 1 | 1 | NA | 1 | 0 | NA | 3 | 0 | NA | 1 | 0 | NA
Dizziness (Nervous system disorders) | 3 | 0 | NA | 2 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 1 | 0 | NA
Headache (Nervous system disorders) | 3 | 0 | NA | 5 | 0 | NA | 2 | 0 | NA | 4 | 0 | NA | 2 | 0 | NA
Paraesthesia (Nervous system disorders) | 1 | 0 | NA | 1 | 0 | NA | 0 | 1 | NA | 3 | 0 | NA | 2 | 0 | NA
Insomnia (Psychiatric disorders) | 2 | 0 | NA | 0 | 0 | NA | 1 | 0 | NA | 4 | 0 | NA | 1 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA | 8 | 0 | NA | 2 | 0 | NA | 8 | 1 | NA | 0 | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | 6 | 0 | NA | 8 | 0 | NA | 4 | 1 | NA | 0 | 0 | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | NA | 1 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0 | NA | 6 | 0 | NA | 3 | 0 | NA | 8 | 1 | NA | 3 | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | NA | 8 | 0 | NA | 3 | 0 | NA | 4 | 1 | NA | 0 | 0 | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 4 | 0 | NA | 0 | 0 | NA | 2 | 0 | NA | 2 | 0 | NA | 2 | 0 | NA
Hypertension (Vascular disorders) | 1 | 0 | NA | 0 | 0 | NA | 0 | 0 | NA | 3 | 0 | NA | 0 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT03484923/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03484923/SAP_001.pdf